CLINICAL TRIAL: NCT05848297
Title: Automated Robotic TCD in Traumatic Brain Injury (ART-TBI)
Brief Title: Automated Robotic TCD in Traumatic Brain Injury
Acronym: ART-TBI
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Wake Forest University (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: HM20026297
Record Dates: First submitted 2023-03-29; First posted 2023-05-08 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Prolonged automated TCD
  Interventions: Device: Transcranial Doppler ultrasonography (TCD)

INTERVENTIONS:
Device: Transcranial Doppler ultrasonography (TCD) — Portable, bedside, non-invasive diagnostic tool used for real-time assessment of cerebral hemodynamics

SUMMARY:
This study's objective is to determine the safety, feasibility and efficacy of prolonged automated robotic TCD monitoring in critically ill patients with severe TBI across multiple clinical sites with varying levels of TCD availability and experience

DETAILED DESCRIPTION:
Upon informed consent, patients will undergo daily automated robotic TCD monitoring sessions for up to 4 hours a day for a total duration of at least 3 days and up to 5 days whenever clinically feasible. TCD monitoring of bilateral middle cerebral artery cerebral blood flow velocity (MCA CBFV) will be performed using a robotic TCD system equipped with bilateral 2-MHz Doppler probes. This system allows for continuous bilateral extended duration recording of MCA CBFV, using robotically controlled TCD probes that allow automated angle correction to maintain optimal MCA insonation.

Safety measures: patient discomfort, device dislodgement or skin lesion at the site of insonation Feasibility: feasibility of using bilateral automated robotic TCD monitoring device on severe TBI patients for >= 4 hrs per day that can provide clinically useful/meaningful data for over 50% of the total monitoring period

Additionally, a 5-question provider survey will be administered at each participating site to obtain bedside nurse and clinician feedback on the perceived safety and feasibility of protocol implementation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18
* Blunt TBI with Glasgow Coma Score (GCS) ≤8
* Injury within 72 hours
* Adequate TCD windows
* Ability to obtain informed consent from a Legally Authorized Representative (LAR)

Exclusion Criteria:

* Catastrophic brain injury with grim prognosis (e.g.: GCS 3 with bilateral mid-position pupil)
* C- spine fracture with evidence of spinal cord injury
* Severe skull or scalp injury precluding device placement
* Planned decompressive hemicraniectomy
* Continuous fever for >6 hours at the time of enrollment (despite treatment)
* Lack of TCD window

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe blunt head trauma with GCS ≤8 within 72 hours of brain injury will be included. Unstable patients and those without identifiable TCD windows will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Patient discomfort (per discretion of the bedside nurse) | 2 years
  To evaluate the safety of prolonged automated robotic TCD monitoring in severe TBI population. Bedside nurse will describe
Inadvertent dislodgement of other intracranial monitoring device/s (if present) | 2 years
  To evaluate the safety of prolonged automated robotic TCD monitoring in severe TBI population. Provider filling out form will describe
Skin changes associated with TCD | 2 years
  To evaluate the safety of prolonged automated robotic TCD monitoring in severe TBI population. Provider filling out form will describe
Provider feedback on safety of prolonged automated robotic TCD monitoring in severe TBI population. | 2 years
  A 5-question provider survey will be administered at each participating site to obtain bedside nurse and clinician feedback on the perceived safety of protocol implementation.
Evaluation of adequate temporal windows | 2 years
  To evaluate the feasibility of prolonged automated robotic TCD monitoring in severe TBI population. Provider completing form will describe
Evaluation of adequate insolation of middle cerebral arteries (MCA) | 2 years
  To evaluate the feasibility of prolonged automated robotic TCD monitoring in severe TBI population. Provider completing form will describe
Provider feedback on the feasibility of prolonged automated robotic TCD monitoring in severe TBI population | 2 years
  A 5-question provider survey will be administered at each participating site to obtain bedside nurse and clinician feedback on the perceived feasibility of protocol implementation, as well as other limiting factors. The survey will be in the format of a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Shraddha Mainali, Principal Investigator — Virginia Commonwealth University
Locations (3):
- United States (3):
  - University of California, Davis, Davis, California
  - Wake Forest University, Winston-Salem, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No